CLINICAL TRIAL: NCT01701804
Title: The Effectiveness of Non-surgical Integrative Package on Failed Back Surgery Syndrome : A Multicenter, Prospective, Case Series Observational Study
Brief Title: The Effectiveness of Non-surgical Integrative Package on Failed Back Surgery Syndrome
Status: Completed | Type: Observational
Sponsor: Jaseng Hospital of Korean Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: JS-CT-2011-2
Record Dates: First submitted 2011-10-22; First posted 2012-10-05 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Failed Back Surgery Syndrome
Keywords: Failed Back Surgery Syndrome
MeSH Terms: conditions — Failed Back Surgery Syndrome | interventions — Acupuncture Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- integrative treatment
  Interventions: Drug: Chuna herbal medicine; Procedure: Chuna manual therapy; Procedure: Acupuncture; Procedure: Bee-venom pharmacoacupuncture

INTERVENTIONS:
Drug: Chuna herbal medicine — 120ml of Chuna herbal medicine(Ostericum koreanum, Eucommia ulmoides, Acanthopanax Sessiliflorus, Achyranthes bidentata, Psoralea corylifolia, Peucedanum japonicum, Cibotium barometz, Lycium chinense, Boschniakia rossica, and Cuscuta chinensis) taken twice a day 30 minutes after meals for 16 weeks
Procedure: Chuna manual therapy — A type of Korean spinal manual therapy administered 5~10 minutes at physician's discretion once a week for 16 weeks. Applies mobilization using High-Velocity, Low-Amplitude thrusts to joints slightly beyond the passive ROM and manual force within the passive ROM without thrusts.
  Other Names: Chuna manipulation
Procedure: Acupuncture — Acupuncture using sterilized disposable needles, sized 0.30X40 mm. Needles left for 15~20 minutes, selecting 6 acupoints(both BL23, BL24, BL25) and other acupoints at physician's discretion, using a total of 10~20 acupoints once a week for 16 weeks.
Procedure: Bee-venom pharmacoacupuncture — Bee-venom pharmacoacupuncture using 30G sterilized bee venom. Selecting 6 acupoints(both BL23, BL24, BL25) and other acupoints at physician's discretion, concentration 10,000:1, 0.1 cc per acupoint, total amount injected 1.0 cc/session once a week for 16 weeks.
  Other Names: BV; Bee-venom therapy

SUMMARY:
The purpose of this study is to investigate the effect of a non-surgical integrative package consisting of Chuna herbal medicine, Chuna manual therapy, bee-venom pharmacoacupuncture, acupuncture on failed back surgery syndrome through means of a prospective case series.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the effect of a non-surgical integrative package on failed back surgery syndrome through means of a prospective case series.

After initial screening, treatment will be administered one session a week for 16 weeks. Patients will be followed up at 4 and 8 weeks after conclusion of treatment.

The integrative package used in this study consists of 120ml of Chuna herbal medicine(Ostericum koreanum, Eucommia ulmoides, Acanthopanax Sessiliflorus, Achyranthes bidentata, Psoralea corylifolia, Peucedanum japonicum, Cibotium barometz, Lycium chinense, Boschniakia rossica, and Cuscuta chinensis) and dried extracts in pill form(Cibotium barometz, Atractylodes japonica) taken twice a day 30 minutes after meals, Chuna manual therapy, intermuscular injections of bee-venom pharmacoacupuncture(Select 6 acupoints, concentration 10,000:1, 0.1 cc per acupoint, total amount injected 1.0 cc/session), acupuncture and allow for NSAID intake during the investigational period. The subject is allowed a maximum of 3 pills/day, taken at a minimum of 8 hrs apart. The number of pills taken will be measured at 4 wks after conclusion of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from low back pain and/or leg pain that does not improve or the return of the symptoms within 1 year of spinal surgery
* Low back pain and/or leg pain with duration at least 3 weeks at baseline
* Low back pain and/or leg pain at least 60mm on VAS scale
* Age between 18 and 60
* Given consent to lumbar MRI
* Voluntary participation with written consent given to study consent form
* Given consent to not receive other treatment concerning pain due to spinal disorders during study participation period

Exclusion Criteria:

* Diagnosis of serious disease(s) which are possible causes of back pain such as malignancy, vertebral fracture, spinal infection, inflammatory spondylitis, cauda equina compression, etc.
* Prior diagnosis of other chronic disease(s) which could affect effectiveness or interpretation of treatment results such as cardiovascular disease, diabetic neuropathy, fibromyalgia, rheumatoid arthritis, Alzheimer's disease, epilepsy, etc.
* Progressive neurologic deficit(s) or concurrent severe neurological symptoms
* Unsuitable for or at risk of complications from acupuncture treatment such as patients with clotting disorders, severe diabetes with risk of infection, serious cardiovascular disease, or undergoing anticoagulant treatment, etc.
* Under prescription of corticosteroids, immuno-suppressant drugs, psychiatric medicine, or other medication considered unsuitable for subjects by the researcher
* Experience of gastroenteric complications after taking NSAIDs or currently undergoing treatment for digestive disorders
* During pregnancy or suspected pregnancy
* Subjects considered unsuitable for clinical trial by the researcher

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patient sampling within Failed Back Surgery Syndrome clinic
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
VAS of low back pain | Baseline, 2nd week, 4th week, 6th week, 8th week, 10th week, 12th week, 14th week, 16th week, 24th week
VAS of radiating leg pain | Baseline, 2nd week, 4th week, 6th week, 8th week, 10th week, 12th week, 14th week, 16th week, 24th week

SECONDARY OUTCOMES:
ODI (Oswestry Disability Index) | Baseline, 4th week, 8th week, 12th week, 16th week, 24th week
SF-36 (Quality of Life) | Baseline, 4th week, 8th week, 12th week, 16th week, 24th week
General assessment(patient/doctor) | 16th week, 24th week
  General assessment of improvement by doctor and patient

CONTACTS AND LOCATIONS:
Overall Officials: Joonshik Shin, OMD, Ph.D, Principal Investigator — Jaseng Hospital of Korean Medicine
Locations (2):
- South Korea (2):
  - Jaseng Hospital of Oriental Medicine, Bucheon-si, Gyeonggi Province
  - Jaseng Hospital of Oriental Medicine, Seoul